CLINICAL TRIAL: NCT01994356
Title: Pilot Study of Physician Self-disclosure of Personal Intrauterine Contraceptive Use Versus Usual Counseling
Brief Title: Physician Self Disclosure of IUC Use
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Mya Zapata, Clinical Lecturer, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IUC Disclosure; N014264 (Other Grant/Funding Number: Sociey of Family Planning)
Record Dates: First submitted 2013-11-19; First posted 2013-11-25 (Estimated); Last update posted 2013-11-25 (Estimated); Status verified 2013-11

CONDITIONS: Contraception
Keywords: Contraceptive counseling; Physician self disclosure; Satisfaction; Intrauterine contraceptive use
MeSH Terms: conditions — Personal Satisfaction

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Usual contraceptive counseling (Active Comparator): subjects received usual contraceptive counseling
  Interventions: Behavioral: Usual contraceptive counseling
- Physician self-disclosure of IUC use (Experimental): subjects received usual contraceptive counseling plus intervention which was Physician self-disclosure of personal IUC use during the counseling
  Interventions: Behavioral: Physician self-disclosure of personal IUC use

INTERVENTIONS:
Behavioral: Physician self-disclosure of personal IUC use — Physicians self-disclosed personal intrauterine contraceptive use to subjects in intervention arm of study during contraceptive counseling
  Arms: Physician self-disclosure of IUC use
Behavioral: Usual contraceptive counseling — all subjects recieved usual contraceptive counseling
  Other Names: contraceptive counseling
  Arms: Usual contraceptive counseling

SUMMARY:
As many as one-third of female healthcare providers use intrauterine contraception (IUC), but only about 8 percent of US women overall do. This begs the question: Might physician self-disclosure of personal IUC use increase IUC use among patients? However, the positive or negative impact of physician self disclosure on IUC uptake or patient satisfaction is generally unknown. The purpose of this study was to evaluate if physician self-disclosure of personal IUC use increases patient use of IUC or impacts patients' satisfaction with their clinical encounter.

DETAILED DESCRIPTION:
We performed a prospective randomized block design pilot trail of usual contraceptive counseling versus usual counseling plus physician self-disclosure of personal intrauterine contraceptive use.

ELIGIBILITY:
Inclusion Criteria:

* reproductive age
* currently sexually active
* scheduled for benign gynecology visit, annual exam, or family planning visit

Exclusion Criteria:

* seeking pregnancy within 1 year
* currently using IUC
* prior sterilization procedure
* currently pregnant

Ages: 18 Years to 44 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 132 (Actual)
Dates: Start 2011-01; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Intrauterine contraceptive use | immediately following clinical encounter and at 2 months
  All subjects were surveyed to determine use of intrauterine contraceptive immediately after their clinical visit where contraceptive counseling was received and at 2 months after their clinical encounter to assess intrauterine contraceptive use.

SECONDARY OUTCOMES:
Satisfaction with clinical encounter | immediately following clinical encounter and at 2 months
  All subjects were surveyed to determine their with satisfaction with their overall clinical encounter immediately following their clinical encounter at at 2 months. Satisfaction was measured using a 5 point scale.

OTHER OUTCOMES:
Satisfaction with contraceptive method | immediately following clinical enocunter and at 2 months
  All subjects were surveyed to determine satisfaction with their contraceptive method of choice immediately following their clinical encounter and at 2 months. Satisfaction was measured using a 5 point scale.
Satisfaction with provider | immediately following clinical encounter and at 2 months
  All subjects were surveyed to determine satisfaction with their provider immediately following their clinical encounter and at 2 months. Satisfaction was measured using a 5 point scale.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Michigan Medical Center, Ann Arbor, Michigan, United States